CLINICAL TRIAL: NCT06727838
Title: A Single-center, Open-label, Fixed-sequence, Self-controlled Pharmacokinetics Study of Metformin and HRS-7535 in Healthy Subjects
Brief Title: Study on Drug Interaction of Metformin Tablets and HRS-7535 Tablets in Healthy Human
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-7535-108
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: HRS-7535 tablets; Drug: Metformin Hydrochloride Extended-release Tablets; Drug: Metformin Hydrochloride Tablets

INTERVENTIONS:
Drug: HRS-7535 tablets — HRS-7535 tablets.
Drug: Metformin Hydrochloride Extended-release Tablets — Metformin Hydrochloride Extended-release Tablets.
Drug: Metformin Hydrochloride Tablets — Metformin Hydrochloride Tablets.

SUMMARY:
This study was a single-center, open, fixed-sequence, self-controlled trial design conducted in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign informed consent before the start of activities related to this experiment, be able to communicate well with the investigators, understand the procedures and methods of this experiment, and be willing to strictly follow the clinical trial protocol to complete this experiment;
2. Healthy male aged 18-50 years old (including both ends of the value, subject to the signing of the informed consent);
3. Weight ≥ 50 kg, and body mass index (BMI): 22~26 kg/m2 (including both ends of the value);
4. Signed informed consent to have no birth plan for 6 months after the last dose, and agreed to take effective contraceptive measures.

Exclusion Criteria:

1. Have a history of drug or food allergy, or are allergic;
2. Inability to swallow, chronic diarrhea and intestinal obstruction, or the presence of multiple other factors affecting the administration and absorption of drugs;
3. QTcF > 450 ms was detected by 12-lead electrocardiogram during screening or there were other abnormalities that were clinically significant as determined by the investigator;
4. Hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, syphilis antibody test positive;
5. Those who smoked more than 5 cigarettes per day in the 3 months prior to screening and could not stop using any tobacco products during the test;
6. Regular drinkers in the 6 months prior to screening, i.e. those who drink more than 14 units of alcohol per week (1 unit = 285 mL for beer, or 25 mL for spirits, or 100 mL for wine) and cannot stop using any alcohol-containing products during the test period, who test positive for alcohol breath test;
7. Patients with a history of drug abuse, drug dependence (consultation) or positive urine drug abuse screening before drug administration;
8. Patients who have received any surgery within 6 months before screening;
9. Participants who have participated in clinical trials of any drug or medical device within 3 months prior to screening (subject to receiving experimental drugs or medical device intervention);
10. Blood donation (or blood loss) and blood donation (or blood loss) ≥ 400 mL within 3 months before screening, or receiving blood transfusion;
11. Patients who had any clinically significant acute disease within 1 month before screening;
12. People who have taken any prescription, over-the-counter, Chinese herbal or health product within 14 days prior to taking the study drug, and plan to take any drug or health product other than the study drug during the trial;
13. Patients with a history of severe hypoglycemia;
14. People with a history of recurrent urinary tract infections, diabetes insipidus or/and genital fungal infections;
15. Previous history of clinical gastric emptance abnormalities (such as gastric outlet obstruction), severe chronic gastrointestinal diseases (such as inflammatory bowel disease, active ulcers);
16. Previous history or family history of medullary thyroid cancer, multiple endocrine adenomatosis type 2, previous history of pancreatitis or symptomatic gallbladder disease;
17. 48h before the first dose until the end of the study, subjects refused to stop drinking or eating foods with high methylxanthine content, such as coffee, tea, cola, chocolate, etc.; For 7 days prior to the first dose until the end of the study, subjects refused to discontinue any beverage or food containing grapefruit; Those who have special dietary requirements and cannot comply with a unified diet;
18. Physical examination, vital signs, laboratory examination, abdominal ultrasound, chest film and other abnormal and clinically significant examination results;
19. Persons who have been vaccinated within 1 month prior to screening or plan to be vaccinated during the trial period;
20. Subjects with other factors deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 0 hour to 24 hours after the last dosing.
Area under the plasma concentration-time curve from time zero to the time of last quantifiable analyte concentration (AUC0-t) | 0 hour to 24 hours after the last dosing.
Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-∞) | 0 hour to 24 hours after the last dosing.

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration (Tmax) | 0 hour to 24 hours after the last dosing.
Terminal half-life ( t1/2) | 0 hour to 24 hours after the last dosing.
Apparent clearance (CL/F) | 0 hour to 24 hours after the last dosing.
Apparent volume of distribution (Vz/F) | 0 hour to 24 hours after the last dosing.
Incidence and severity of adverse events (AEs) | 0 hour to 24 hours after the last dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided